CLINICAL TRIAL: NCT01346371
Title: The Effect of BEPREVE (Bepotastine Besilate Ophthalmic Solution) 1.5% on Tear Film Osmolarity and Tear Film Lipid Layer
Brief Title: The Effect of BEPREVE 1.5% on Tear Film Osmolarity and Tear Film Lipid Layer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minnesota Eye Consultants, P.A. (Industry)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAC-01-11
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic; conjunctivitis; Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic; Conjunctivitis | interventions — Lubricant Eye Drops; bepotastine besilate; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Refresh Tears® eye drops (Placebo Comparator): Must add drops twice a day every day during trial enrollment.
  Interventions: Drug: Bepreve 1.5% Ophthalmic Solution
- Bepreve® 1.5% solution (Experimental): Must add drops twice a day every day while enrolled in trial.
  Interventions: Drug: Refresh Tears 0.5% Lubricant Eye Drops

INTERVENTIONS:
Drug: Refresh Tears 0.5% Lubricant Eye Drops
  Arms: Bepreve® 1.5% solution
Drug: Bepreve 1.5% Ophthalmic Solution
  Arms: Refresh Tears® eye drops

SUMMARY:
The purpose of this study is to compare the effect of Bepreve® with an artificial-tear eye drop on the quality of your tears.

DETAILED DESCRIPTION:
This is a single-center, randomized, parallel group, placebo-controlled study to evaluate the effect of BEPREVE compared to a placebo eye drop on the measurement of tear film osmolarity and tear film lipid layer in patients with allergic conjunctivitis.

Subjects will be screened for this study on day one of dosing with the test article. Subjects who sign the informed consent form and who meet all inclusion/exclusion criteria will be eligible for participation in this study. They will be assigned sequentially, according to a computer generated randomization list, in a ratio of 1:1 to receive either BEPREVE™ (bepotastine besilate ophthalmic solution) 1.5% or REFRESH TEARS® Lubricant Eye Drops (1:1). Subjects will instill one drop of test article either BEPREVE™ or REFRESH TEARS® into the study eyes twice daily for a maximum of 60 days. Subjects will be seen for evaluation on Days 0, 28±3, and 56±3 following randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female at least 18 years of age who are diagnosed with allergic conjunctivitis.
2. Have documented positive skin prick puncture test to at least one (1) seasonal allergen (e.g., grasses, trees, weeds, or other allergens) within two (2) years of Visit 1.
3. Agree not to have any other ocular drops in study eyes within 2 days prior to the initiation of dosing with the test article or throughout the duration of the study.
4. Have a Best Corrected Visual Acuity of 20/200 or better in either eye.
5. Are willing/able to follow instructions from the study investigator and his/her staff.
6. Be willing/able to return for all required study visits, to follow instructions from the study investigator and his/her staff.
7. Are able to self-administer test article (or have a caregiver available to instill all doses of test article).
8. Have signed informed consent approved by Institutional Review Board or Independent Ethics Committee.

Exclusion Criteria:

1. Have known hypersensitivity to either BEPREVE™ or REFRESH TEARS® or to any component of the test article (including "procedural" medications such as anesthetic and/or fluorescein drops, dilating drops, etc.).
2. Have active corneal pathology noted in the study eye at the screening visit. Active corneal pathology is defined as corneal pathology that is non-stable, or greater than mild, or will compromise assessment of the safety or efficacy of treatment.
3. Have used topical, ocular, inhaled or systemic steroids within 14 days prior to screening.
4. Have a history of abuse of alcohol/drugs within six months prior to the screening visit.
5. Are pregnant or nursing/lactating.
6. Have participated in any other study of an investigational drug or device within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Fahmy, O.D., Principal Investigator — Minnesota Eye Consultants
Locations (1):
- Minnesota Eye Consultants, P.A., Minneapolis, Minnesota, United States

REFERENCES:
- See also: Minnesota Eye Consultants — http://www.mneye.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began Aug 15, 2011 and concluded June 11, 2012. There are a variety of sources we recruited our subjects from which is outlined below:
  Email. PI referrals, employee, and subject referrals. Flyers posted around college campuses. Website clinicaltrial.gov.
Period: Overall Study
Arm/Group | Refresh Tears® Eye Drops | Bepreve® 1.5% Solution
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Refresh Tears® Eye Drops | Bepreve® 1.5% Solution | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (13) | 35 (12) | 38 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Tear Osmolarity
Description: The TearLab Osmolarity System will be used to assess tear film osmolarity, measured in mOsms/L.
Time Frame: 56 days after initial screening visit
Population: Analysis per protocol as ITT and LOCF for all subject eyes.
Measure: Mean (Standard Deviation); unit: mOsM/L
Units Other Than Participants: Eyes
Arm/Group | Refresh Tears® Eye Drops | Bepreve® 1.5% Solution
Number analyzed (Participants) | 20 | 20
Number analyzed (Eyes) | 40 | 40
mOsM/L | 303 (3.13) | 303 (2.57)

ADVERSE EVENTS:
Arm/Group | Refresh Tears® Eye Drops | Bepreve® 1.5% Solution
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 10/20 | 14/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refresh Tears® Eye Drops (N=20) | Bepreve® 1.5% Solution (N=20)
Ocular Irritation (Eye disorders) | 2 (2) | 1 (1)
Ocular Burning (Eye disorders) | 5 (5) | 4 (4)
Ocular itching (Eye disorders) | 8 (9) | 7 (7)
Cold like symptoms (General disorders) | 7 (7) | 4 (5)
Stomach problems (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bad Taste in mouth (General disorders) | 0 (0) | 7 (7)
General eye discomfort (Eye disorders) | 1 (2) | 1 (3)
Joint/muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No